CLINICAL TRIAL: NCT03508986
Title: The Chinese Familial Parkinson's Disease Registry
Brief Title: Chinese FPD Registry
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: CFPDR
Record Dates: First submitted 2018-04-11; First posted 2018-04-26 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extraction of DNA from peripheral blood of patients and other family members in familial PD
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the Chinese Familial Parkinson's disease Registry (CFPDR) is to develop a database of patients with familial Parkinson's disease (PD) in China.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common disorder among degenerative neurological disease. Familial PD (FPD) has its unique clinical feature and genetic basis. We aim to establish a database of FPD,and characterize the clinical feature, genetic basis, environmental factors and their interactions FPD in China.

Method:

1. Clinical feature will be measured by scales and neurological tests.Standard scales includes: Unified Parkinson's Disease Rating Scale(UPDRS), Hoehn-Yahr stages, NMSS, MMSE, PDSS(Parkinson disease sleep scales),Rapid Eye Movement Sleep Behaviour Disorder Questionnaire(RBDQ-HK),ESS(Epworth Sleepiness Scale),Rome III functional constipation scale，SCOPA-AUT (the Scale for Outcomes in PD for Autonomic Symptoms)，PFS(Parkinson Fatigue Scale)，CH-RLSq，Hyposmia rating scale(HRS)HAMILT depression scale，the 39-item Parkinson's Disease Questionnaire(PDQ-39)，Freezing of gait scale(FOG)，dyskinesia related scales, Wearing-off scale(WO)
2. Peripheral blood from patients and other members in family will be collected for familial PD genetic testing.
3. The environmental factors are exploded by questionnaires including smoking,drinking, pesticide and heavy metals.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease, and either family history of Parkinson's disease (first or second degree family member affected by Parkinson's disease) AND/OR Clinical diagnosis of Parkinson's disease and their parents are close relatives(First or second degree family member of an Index Case, affected or unaffected by Parkinson's disease).

Exclusion Criteria:

* Lack of capacity to consent to participate in the project

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients in hospitals or community
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Database of Familial Parkinson's disease | 10 years
  To collect 1500 patients with familial Parkinson's disease and establish the database of Familial Parkinson's disease (FPD) in mainland China.
Risk Factors | 10 years
  To characterize clinical feature and environmental factors among Chinese familial parkinson's disease
Genetic Basis | 10 years
  To characterize the genetic basis of Chinese FPD and detect clinically relevant genetic variants in these cases

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

REFERENCES:
- [Background] Yan W, Tang B, Zhou X, Lei L, Li K, Sun Q, Xu Q, Yan X, Guo J, Liu Z. TMEM230 mutation analysis in Parkinson's disease in a Chinese population. Neurobiol Aging. 2017 Jan;49:219.e1-219.e3. doi: 10.1016/j.neurobiolaging.2016.10.007. Epub 2016 Oct 11. PMID 27814995
- [Background] Yang Y, Tang BS, Weng L, Li N, Shen L, Wang J, Zuo CT, Yan XX, Xia K, Guo JF. Genetic Identification Is Critical for the Diagnosis of Parkinsonism: A Chinese Pedigree with Early Onset of Parkinsonism. PLoS One. 2015 Aug 21;10(8):e0136245. doi: 10.1371/journal.pone.0136245. eCollection 2015. PMID 26295349
- [Background] Li K, Tang BS, Liu ZH, Kang JF, Zhang Y, Shen L, Li N, Yan XX, Xia K, Guo JF. LRRK2 A419V variant is a risk factor for Parkinson's disease in Asian population. Neurobiol Aging. 2015 Oct;36(10):2908.e11-5. doi: 10.1016/j.neurobiolaging.2015.07.012. Epub 2015 Jul 11. PMID 26234753
- [Result] Liu Z, Guo J, Li K, Qin L, Kang J, Shu L, Zhang Y, Wei Y, Yang N, Luo Y, Sun Q, Xu Q, Yan X, Tang B. Mutation analysis of CHCHD2 gene in Chinese familial Parkinson's disease. Neurobiol Aging. 2015 Nov;36(11):3117.e7-3117.e8. doi: 10.1016/j.neurobiolaging.2015.08.010. Epub 2015 Aug 15. PMID 26343503
- [Result] Guo JF, Li K, Yu RL, Sun QY, Wang L, Yao LY, Hu YC, Lv ZY, Luo LZ, Shen L, Jiang H, Yan XX, Pan Q, Xia K, Tang BS. Polygenic determinants of Parkinson's disease in a Chinese population. Neurobiol Aging. 2015 Apr;36(4):1765.e1-1765.e6. doi: 10.1016/j.neurobiolaging.2014.12.030. Epub 2015 Jan 6. PMID 25623333